CLINICAL TRIAL: NCT01997164
Title: An Open-Label, Dose-Escalation Study of the Safety and Tolerability of Intravitreal (IVT) REGN910-3 and IVT REGN910 in Patients With Either Neovascular AMD or DME
Brief Title: Study of Intravitreal (IVT) REGN910-3 and IVT REGN910 in Patients With Either Neovascular ("Wet") Age Related Macular Degeneration (AMD) or Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R910-3-OD-1403
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Neovascular Age-Related Macular Degeneration; Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohorts 1 through 4 (Experimental): Participants in cohorts 1 through 4 will receive IVT REGN910-3 and IAI
  Interventions: Drug: REGN910-3; Drug: Intravitreal Aflibercept Injection (IAI)
- Cohort 5 (Experimental): Participants in cohort 5 will receive IVT REGN910 and IAI
  Interventions: Drug: REGN910; Drug: Intravitreal Aflibercept Injection (IAI)

INTERVENTIONS:
Drug: REGN910-3
  Arms: Cohorts 1 through 4
Drug: REGN910
  Arms: Cohort 5
Drug: Intravitreal Aflibercept Injection (IAI)
  Other Names: EYLEA®

SUMMARY:
The primary objective of the study is to investigate the safety and tolerability of intravitreal (IVT) REGN910-3 and IVT REGN910 in patients with neovascular age-related macular degeneration (AMD), and separately in patients with diabetic macular edema (DME).

ELIGIBILITY:
Key Inclusion Criteria:

1. For patients with AMD:

   1. Active subfoveal choroidal neovascularization (CNV) secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by FA or OCT in the study eye, as determined by the investigator
   2. Men or women ≥50 years and older
2. For patients with DME:

   1. Patients with clinically significant DME with central involvement (≥300 μm in the central subfield on spectral domain OCT)
   2. Men or women ≥18 years and older

Key Exclusion Criteria:

1. For patients with neovascular AMD:

   1. Evidence of choroidal neovascularization (CNV) due to any cause other than AMD in either eye
   2. Evidence of diabetic retinopathy (DR) or DME in either eye
2. For patients with DME: Evidence of neovascular AMD or CNV due to any cause in either eye
3. Prior IAI in either eye
4. IVT bevacizumab, ranibizumab, or pegaptanib sodium in the study eye within 8 weeks of day 1 or an AE with any of these previous treatments that would preclude administration of drug in this study
5. Any prior treatment with angiopoietin inhibitors
6. Any prior systemic (IV) anti-VEGF administration
7. History of vitreoretinal surgery in the study eye
8. Pan retinal laser photocoagulation or macular laser photocoagulation in the study eye within 3 months of the screening visit
9. Previous use of intraocular or periocular corticosteroids in the study eye within 4 months of screening

(The inclusion/ exclusion criteria provided above are not intended to contain all considerations relevant to a subject's potential participation in this clinical trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Change from baseline to week 24
  Incidence of TEAEs through week 24 in patients treated with IVT REGN910-3 and IVT REGN910 TEAEs through week 24 in patients treated with IVT REGN910-3 and IVT REGN910

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile | Baseline to week 24
  PK profile may include, but is not limited to, the following:
  * AUCall - area under the curve (AUC) computed from time zero to the time of the last concentration
  * AUCall/Dose - AUCall-to-dose ratio
  * AUClast - AUC computed from time zero to the time of the last positive concentration
  * AUClast/Dose - AUClast-to-dose ratio
  * Cmax - the peak concentration
  * Cmax/Dose - Cmax-to-dose ratio
Development of Anti-drug antibodies (ADA) after IVT injection of REGN910-3 | Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- United States (5):
  - Beverly Hills, California
  - Winter Haven, Florida
  - Boston, Massachusetts
  - West Columbia, South Carolina
  - Abilene, Texas